CLINICAL TRIAL: NCT02635412
Title: Delivery Timing in Morbidly Adherent Placentas: a Randomized, Controlled Trial
Acronym: MAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Never approved by the IRB
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-MS-16-0085
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Morbidly Adherent Placenta; Placenta Accreta
Keywords: Placenta; Accreta; Morbidly; Adherent Placenta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Scheduled delivery at 34 weeks (Placebo Comparator): Scheduled delivery at 34 weeks (range 33 weeks 5 days to 34 weeks 3 days)
  Interventions: Other: Scheduled timing of delivery
- Scheduled delivery at 36 weeks (Active Comparator): Scheduled delivery at 36 weeks (range 35 weeks 5 days to 36 weeks 3 days)
  Interventions: Other: Scheduled timing of delivery

INTERVENTIONS:
Other: Scheduled timing of delivery

SUMMARY:
This is a randomized controlled trial to investigate the optimal timing of delivery in clinically stable women with a suspected morbidly adherent placenta.

DETAILED DESCRIPTION:
This is a randomized controlled trial to investigate the optimal timing of delivery in clinically stable women with a suspected morbidly adherent placenta dispositioned for a scheduled delivery. The primary outcome will be assessed by comparing the composite neonatal morbidity and composite maternal morbidity between the two groups (delivery at 34 versus 36 weeks gestational age).

ELIGIBILITY:
Inclusion Criteria:

* Women with monographically morbidly adherent placenta with or without a placenta previa.
* Scheduled delivery via cesarean hysterectomy

Exclusion Criteria:

* Delivery planned prior to 36 weeks (e.g. non-reassuring fetal status, preterm labor, severe preeclampsia, other medical/fetal indication for delivery as determined by the managing physician).

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Composite neonatal morbidity | Within 72 hours of newborn discharge
Maternal neonatal morbidity | Within 72 hours of patient discharge